CLINICAL TRIAL: NCT01202240
Title: A Phase 1, Open Label, Fixed-Sequence Study To Estimate The Effect Of Ketoconazole On The Pharmacokinetics Of Tasocitinib (CP-690,550) In Healthy Volunteers
Brief Title: Effect Of Ketoconazole On The Pharmacokinetics Of Tasocitinib (CP-690,550) In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3921054
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Drug-Drug Interaction; Healthy Volunteers; Tasocitinib (CP-690; 550); Ketoconazole
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tasocitinib (CP-690,550) plus Ketoconazole (Experimental)
  Interventions: Drug: Tasocitinib (CP-690,55) plus Ketoconazole

INTERVENTIONS:
Drug: Tasocitinib (CP-690,55) plus Ketoconazole — Period 1, Day 1: tasocitinib (CP-690,550) as a single oral 10 mg dose given as two 5 mg tablets Period 2, Days 1-2: ketoconazole as a daily single oral 400 mg (dose given as two 200 mg tablets Period 2, Day 3: ketoconazole as a single oral 400 mg dose given as two 200 mg tablets PLUS tasocitinib (CP-690,550) as a single oral 10 mg oral dose given as two 5 mg tablets Period 2, Day 4: No treatment (discharge)

SUMMARY:
Estimate the effect of oral ketoconazole administration (400 mg once daily over 3 days) on the pharmacokinetics (process by which the drug is absorbed, distributed, metabolized, and eliminated by the body) of single 10 mg dose of tasocitinib (CP-690,550) in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 18 and 55 years

Exclusion Criteria:

* Clinically significant disease
* Recent history of serious infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
AUCinf of tasocitinib (CP-690,550) | 5 days

SECONDARY OUTCOMES:
AUClast, Cmax, and Tmax of tasocitinib (CP-690,550) | 5 days
Safety: laboratory tests, AE reporting and vital signs | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- [Derived] Gupta P, Chow V, Wang R, Kaplan I, Chan G, Alvey C, Ni G, Ndongo MN, LaBadie RR, Krishnaswami S. Evaluation of the effect of fluconazole and ketoconazole on the pharmacokinetics of tofacitinib in healthy adult subjects. Clin Pharmacol Drug Dev. 2014 Jan;3(1):72-7. doi: 10.1002/cpdd.71. Epub 2013 Oct 8. PMID 27128233
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921054&StudyName=Effect%20Of%20Ketoconazole%20On%20The%20Pharmacokinetics%20Of%20Tasocitinib%20%28CP-690%2C550%29%20In%20Healthy%20Volunteers